CLINICAL TRIAL: NCT01379352
Title: Vecuronium Requirements According to the Operation Phase During Liver Transplantation Under Desflurane Anesthesia
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Gaab Soo Kim, Professor, Samsung Medical Center
Other Study IDs: 2011-04-015
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Liver Transplantation
Keywords: liver transplantation; vecuronium

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High MELD group: Preoperative MELD score greater than 20
- Low MELD group: Preoperative MELD score lesser than 20

SUMMARY:
The vecuronium requirements may be reduced for recipients of living donor liver transplantation, as the vecuronium is eliminated principally by the liver. Furthermore, the requirements may be different according to the phase of surgery. The requirements may also be different according to the preoperative hepatic function as measured by MELD score during prehepatic phase, or graft to recipient body weight ratio (GRWR) during neohepatic phase. Therefore, the investigators are trying to investigate the difference of vecuronium requirements according to the phase of surgery or MELD score, GRWR.

DETAILED DESCRIPTION:
The vecuronium requirements may be reduced for recipients of living donor liver transplantation, as the vecuronium is eliminated principally by the liver. Furthermore, the requirements may be different according to the phase of surgery. The requirements may by further reduced during anhepatic phase of liver transplantation. And the requirements may be increased as the graft functions during neohepatic phase.

We also postulated that the requirements may be different according to the preoperative hepatic function during preanhepatic phase, and according to the graft to recipient body weight ratio (GRWR) during neohepatic phase.

Therefore, we are trying to investigate the difference of vecuronium requirements according to the phase of surgery, MELD score, GRWR.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective living donor liver transplantation

Exclusion Criteria:

* patients who can not undergo train-of-four test due to central or peripheral neuromuscular disease.
* patients with severe cardiopulmonary diseases.
* patients who received transfusion with more than 10 units of packed red blood cells.
* primary non-functioning graft immediately after reperfusion of the graft.
* patients who administered drugs that influences the metabolism of vecuronium (such as anticonvulsant: phenytoin, carbamazepine, primidone, sodium valproate)
* patients undergoing cadaver donor liver transplantation

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective living donor liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
vecuronium requirements during preanhepatic phase | during prehepatic phase of liver transplantation
  total vecuronium requirements as guided by Train-of-four neuromuscular monitoring during preanhepatic phase
vecuronium requirements during anhepatic phase | during anhepatic phase of liver transplantation
  total vecuronium requirements as guided by Train-of-four neuromuscular monitoring during anhepatic phase
vecuronium requirements during neohepatic phase | during neohepatic phase of liver transplantation
  total vecuronium requirements as guided by Train-of-four neuromuscular monitoring during neohepatic phase

CONTACTS AND LOCATIONS:
Overall Officials: Gaab Soo Kim, M.D.,Ph.D., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea